CLINICAL TRIAL: NCT02543307
Title: Quality and Process Improvement Using Nurse-led Patient Pathways in an Orthopedic Hospital
Brief Title: Effects of Nurse-led Patient Pathways
Acronym: NPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Balgrist University Hospital (Other); Ebnet-Foundation (Unknown); Swiss Association Balgrist (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Lorenz Imhof, Prof. Dr., Zurich University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P270248_151704; 2011_0248 (Other: KEK_ZH-ID)
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Musculoskeletal Diseases
Keywords: Hip Replacement; Spinal Diseases; Rotator Cuff Reconstruction; Nursing; Nurse-led; Pathways; Patient Satisfaction; Quality of Nursing Care
MeSH Terms: conditions — Musculoskeletal Diseases; Spinal Diseases; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse-led Patient Pathways (Experimental): Patients were cared for under the three NPP developed for the orthopedic populations: NPP-1) patients with total hip arthroplasty; NPP-2) exploration and decompression of the spinal cord; and NPP-3) rotator cuff reconstruction. NPP are characterized by four principles: evidence-based nursing, patient and family centred care, comprehensive discharge planning beyond hospital discharge and nurses' responsibility for patients' processes. The principles support and strengthen patient and family preferences as well as formalize nursing activities, and therefore contribute to process transparency in relation to other health care professionals. Aims: to improve patients' and health care professionals' as well as institutional outcomes.
  Interventions: Procedure: Nurse-led Patient Pathways
- Standard usual nursing care (No Intervention): Patients in the control group will receive usual nursing care, which is based on the institutional principles and standards of care for surgical patients. Based on the type of surgery and assessment of the nurse the nursing process is used to care for the patients. The nurses will be ending their activities with discharge of the patients.

INTERVENTIONS:
Procedure: Nurse-led Patient Pathways — The NPP include a comprehensive needs and goal assessment. Patients appreciated written information provided at an early stage of their hospital stay that helped to prepare them for discharge. The NPP continue with pre- and post-operative patient care, and conclude with a newly implemented follow-up phone call after hospital discharge. Nursing interventions were presented in a checklist format, based on scientific and clinical evidence. The NPP were developed with regard to patient and family centered goals and objectives and were explicitly emphasized in the NPP. NPP guided the nursing care plan. Nurses act as advocates for patients' interests. Therefore NPPs represent a means to formalize these nursing activities and contribute to transparency in relation to other health professionals.
  Arms: Nurse-led Patient Pathways

SUMMARY:
Objectives: This quasi-experimental pre-post-study investigated the effect of newly developed Nurse-led Patient Pathways (NPP) designed to improve patients', and health care professionals' as well as institutional outcomes.

Intervention: In the IG patients were cared for under the three newly developed NPP. NPP are characterized by four principles: evidence-based nursing, patient and family centered care, comprehensive discharge planning beyond hospital discharge and nurses' responsibility for patients' processes. The principles support and strengthen patient and family preferences as well as formalize nursing activities, and therefore contribute to process transparency in relation to other health care professionals.

Outcomes: Primary Outcomes were defined as quality of nursing care (nursing care index, NCI), and patient satisfaction (patient satisfaction with nursing care quality, PSNCQ). Secondary outcomes were defined as 1) nursing work environment (nursing work index revised, NWI-R; and nursing workplace quality, NWQ), and 2) institutional-related costs (length of hospital stay, LOS; nursing time and nursing costs). Additionally, nurses' and other health care professionals' experiences of intervention translation will be explored.

DETAILED DESCRIPTION:
In Switzerland, the hospitalization rate of patients with musculoskeletal disorders has increased within the last decade. For example, recent data shows that Switzerland had the highest rate of hip replacement surgery in Europe. Due to the introduction of diagnosis related groups in Switzerland, there is increased pressure to reduce length of hospital stay and increase economic efficiency.

To achieve the required economic efficiency, there is a trend towards standardization of care delivery processes, often in the form of care pathways. The European Pathway Association has defined care pathways as a complex intervention. Pathways should incorporate evidence based care, best practices and patient expectations. As such, care pathways depend on communication and coordination between team members, patients and families, as well as defined roles and sequenced activities.

However, care pathways are often criticized for their organization-driven focus, the lack of a patient centered perspective or missing a holistic approach to care. Therefore, the Balgrist University Hospital and the Zurich University of Applied Sciences developed NPP to enhance patients', and health care professionals' as well as institutional outcomes.

Method: A quasi-experimental prospective study with a pre-post sample design will be conducted. Usual care will be given in the control group (Pre) and compared with a group of patients that were assigned to NPP (Post). The study will be conducted on the two largest orthopedic units at the Balgrist University Hospital, a highly specialized center in musculoskeletal care, located in the Canton of Zurich.

1. A convenience sample will be recruited, consisting of 558 surgical patients hospitalized for total hip arthroplasty, exploration and decompression of the spinal cord, and rotator cuff reconstruction. Demographic, clinical data as well as data to measure quality of nursing care, patient satisfaction, and costs will be obtained,
2. A sample of 38 nurses will be recruited, which are working on the two units. Demographic data and data to measure nursing work environment will be contained,
3. Additionally, a sample of 6 nurses and 5 other health care professionals' (directly involved in patients care) will be recruited to explore experiences of intervention translation within 2 focus group sessions.

The quantitative data analyses will be performed using statistical tests appropriate to the sample size, measurement level, distribution and the independence of variables. For group control appropriate tests for independent groups were used in respect to provision of necessary assumptions. Statistically significance was set on Alpha .05 with undirected hypothesis testing, if necessary correction for multiple testing will be included. Qualitative data analysis will be performed using content analysis.

We hypothesized that the NPP-group (post) will be experienced higher quality of nursing care and increased patient satisfaction, without an increase in health care costs. Secondary outcomes will be enhanced work environment for the nurses.

ELIGIBILITY:
1. patients

   Inclusion Criteria:
   * surgical patients hospitalized for total hip arthroplasty, exploration and decompression of the spinal cord, and rotator cuff reconstruction,
   * age 18 years or older,
   * German speaking (oral and written),
   * consents to the use of patient data (chart review),
   * give informed consent (patient survey)

   Exclusion Criteria:
   * inclusion criteria will be not met
   * patients that had cognitive deficits such that they were unable to provide informed consent
2. nurses (survey and interview)

   Inclusion Criteria:
   * age 18 years or older,
   * works on one of the two study units
   * give informed consent

   Exclusion Criteria:

   - inclusion criteria will be not met
3. other health care professionals

Inclusion Criteria:

* directly involved in patients care
* give informed consent

Exclusion Criteria:

- inclusion criteria will be not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Nursing Care Index (NCI) between pre and post intervention group | Pre-data will be gathered over an eight month period for the control group. After a 4-month break for the implementation of the NPP, the 10-month post-data collection period for the NPP-group will be started.
  The NCI was used to measure the quality of nursing care. The self-developed instrument included 35 items with yes/no-answers for each item. Data will be generated from entries in the patient's electronic clinical record. The total NCI-score was calculated by computing the average value of all mean values of the subscales. NCI-scores could range between zero (lowest quality) and one (highest quality). Six subscales will be used in order to reflect the key principles of NPPs (Initial Pain Assessment, Needs and Goal Assessment, Family Centred Care, Care Planning, Post-surgical Care, Discharge Planning).
Change in Patient Satisfaction with Nursing Care Quality (PSNCQ) between pre and post intervention group | Pre-data will be gathered over an eight month period for the control group. After a 4-month break for the implementation of the NPP, the 10-month post-data collection period for the NPP-group will be started.
  The PSNCQ Questionnaire was used to measure the patient satisfaction with nursing care quality. The 19-item instrument is a validated and common used instrument in clinical settings to measure patient satisfaction. The patients evaluated key areas of nursing care during their hospital stay on a 5-point Likert in terms of whether the quality was excellent (5 points), very good, good, fair or poor (1 point). The maximum value (5) reflected a high level of satisfaction and the lowest value (1) indicated a deep dissatisfaction with the nursing performance. Data were collected using a survey mailed to the patients within the first week after discharge. For the first 84 patients in the control group survey was not possible because data collection took place more than one week after discharge.

SECONDARY OUTCOMES:
Change in nursing work environment (nursing work index revised, NWI-R) between pre and post intervention group | Data will be gathered ones for the control group close before implementation of the NPP, and ones after 8 month of implementation of NPP.
  The NWI-R is a validated and common instrument in clinical settings to measure the quality of nursing work environment. The NWI-R includes 51 items that are rated on a 4-point Likert (strongly agree (4 points), agree, disagree, strongly disagree (1 point). The total NWI-R-score will be calculated by computing the average over all 51 items. NWI-R-scores could range between 0 (dissatisfaction with nursing work environment) and 1 (satisfaction with nursing work environment). Three NWI-R subscales are included (Leadership & Development, Resources & Autonomy, and Cooperation & Competence).
Change in nursing work environment (nursing workplace quality, NWQ) between pre and post intervention group | Data will be gathered ones for the control group close before implementation of the NPP, and ones after 8 month of implementation of NPP.
  The NWQ Questionnaire is a self-developed instrument to measure the quality of nursing work environment in a shorter version, based on characteristics of magnet hospitals. The NWQ Questionnaire includes 8 items that are rated on a visual analog scale (strongly agree (100 points) and strongly disagree (0 points). The total NWQ-score will be calculated by computing the average over all 8 items. NWI-R-scores could range between 0 (dissatisfaction with nursing work environment) and 100 (satisfaction with nursing work environment).
Change in institutional-related costs (length of hospital stay, LOS; nursing time and nursing costs). | Pre-data will be gathered over an eight month period for the control group. After a 4-month break for the implementation of the NPP, the 10-month post-data collection period for the NPP-group will be started.
  Data related to costs were collected using 1) length of stay in days, retrieved from patients' clinical record entries (based on date of admission and date of discharge), 2) nursing time for patient care in minutes, and 3) costs of nursing care per case in Swiss franc (CHF), provided by the comptroller department using data from the LEP® method, a workload measurement system for the healthcare system. Higher values will be indicated higher institutional-related costs.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Imhof, Prof Dr, Principal Investigator — Zurich University of Applied Sciences
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland